CLINICAL TRIAL: NCT04161469
Title: Laser Closure of Anal Fistula (FiLaC); Do we Need to Close Internal Orifice?
Brief Title: Laser Closure of Anal Fistula (FiLaC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Surp Pırgiç Armenian Hospital (Other)
Responsible Party: Principal Investigator, Kursat Serin, Asistant Profesor, Surp Pırgiç Armenian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10
Record Dates: First submitted 2019-10-22; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Anal Fistula; Fistula in Ano; Sphincter Ani Incontinence
Keywords: sphincter injury; anal abscess; incontinence
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: The FiLaC procedure was performed using a ceramic diode laser platform (12 watts, 1470-nm wavelength). The laser fiber was introduced into the fistula tract via the external orifice using the seldinger maneuver until the internal orifice was found. The fiber delivered laser energy homogenously at 3600, causing shrinkage of the fistula tract around the fiber while it was withdrawn at the speed of 1 mm/s (2). We planned to randomized patients in two groups. Group 1) FiLaC closure of the tract, group 2) FiLaC closure of the tract with an additional surgical technique as the closure of the internal orifice with a purse-string suture using 2-0 polyglactin (VicrylR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Patients diagnosed with anal fistula treated by laser closure of the tract
  Interventions: Procedure: Laser closure of the anal fistula tract (FiLaC)
- Group 2 (Other): Patients diagnosed with anal fistula treated by laser closure of the tract with an additional surgical technique as the closure of the internal orifice with a purse-string suture using 2-0 polyglactin
  Interventions: Procedure: Laser closure of the anal fistula tract (FiLaC); Procedure: Internal orifice closure

INTERVENTIONS:
Procedure: Laser closure of the anal fistula tract (FiLaC) — The FiLaC procedure was performed using a ceramic diode laser platform (12 watts, 1470-nm wavelength). The laser fiber was introduced into the fistula tract via the external orifice using the seldinger maneuver until the internal orifice was found. The fiber delivered laser energy homogenously at 3600, causing shrinkage of the fistula tract around the fiber while it was withdrawn at the speed of 1 mm/s
Procedure: Internal orifice closure — Closure of internal orifice with a purse-string suture using 2-0 polyglactin suture material.
  Arms: Group 2

SUMMARY:
Laser closure of the perianal fistula is the minimally invasive and low complication rate procedure which is a life-saving way for complex fistulas, preserving anal sphincter injury. Unfortunately, wide range success rate reported before (30-80%), the investigators are searching to reach better rates. Internal closure of the fistula orifice offered by some authors. The investigators are aimed to identify the efficiency of this.

DETAILED DESCRIPTION:
Despite the developments in the surgical field, the treatment of anal fistula is still a challenging problem, especially in complex, transsphincteric cases. The surgical treatment aims to avoid recurrences and also to preserve normal sphincter functions. The FiLaC procedure was recently reported non-invasive technique in perianal fistulas for treatment and preserving anal sphincter function with a good success rate. In 2018, one of our colleagues published a 40% complete healing rate by using only FiLaC technique in 103 consecutive perianal fistula patients (Prof. Cem Terzi). Some authors advocated that the closure of the internal orifice increasing the success rate. Therefore, the investigators decided to modify the surgical technique focusing closure of the internal opening associated with the FiLaC procedure.

ELIGIBILITY:
Inclusion Criteria:

* complex anal fistula
* high anal fistulas
* recurrent anal fistulas

Exclusion Criteria:

* superficial anal fistulas
* multibranching anal fistulas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from perianal fistula disease severity score at 6 months | 6th month after the surgery
  0: no active disease or complete healing,
  1. slight drainage with minimal symptoms,
  2. persistent symptomatic drainage,
  3. painful symptomatic drainage,
  4. severe perianal disease potentially requiring diversion

CONTACTS AND LOCATIONS:
Locations (1):
- Surp Pırgic AH, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR)

REFERENCES:
- [Result] Terzi MC, Agalar C, Habip S, Canda AE, Arslan NC, Obuz F. Closing Perianal Fistulas Using a Laser: Long-Term Results in 103 Patients. Dis Colon Rectum. 2018 May;61(5):599-603. doi: 10.1097/DCR.0000000000001038. PMID 29528908
- [Result] Wilhelm A. A new technique for sphincter-preserving anal fistula repair using a novel radial emitting laser probe. Tech Coloproctol. 2011 Dec;15(4):445-9. doi: 10.1007/s10151-011-0726-0. Epub 2011 Aug 16. PMID 21845480
- [Result] Ozturk E, Gulcu B. Laser ablation of fistula tract: a sphincter-preserving method for treating fistula-in-ano. Dis Colon Rectum. 2014 Mar;57(3):360-4. doi: 10.1097/DCR.0000000000000067. PMID 24509460
- [Result] Wilhelm A, Fiebig A, Krawczak M. Five years of experience with the FiLaC laser for fistula-in-ano management: long-term follow-up from a single institution. Tech Coloproctol. 2017 Apr;21(4):269-276. doi: 10.1007/s10151-017-1599-7. Epub 2017 Mar 7. PMID 28271331